CLINICAL TRIAL: NCT04962191
Title: Technology Study: Measuring Potential Impact of Research Use Only Rapid EGFR Testing on Standard of Care
Brief Title: Idylla EGFR Lung Trial
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Anthony Magliocco (Industry)
Responsible Party: Sponsor-Investigator, Anthony Magliocco, Principal Investigator, Protean BioDiagnostics
Organization: Protean BioDiagnostics (Industry)
Other Study IDs: R20-00012
Record Dates: First submitted 2020-12-17; First posted 2021-07-14 (Actual); Last update posted 2021-07-14 (Actual); Status verified 2021-07

CONDITIONS: Lung Cancer; Technology; Oncology
Keywords: Protean BioDiagnostics
MeSH Terms: conditions — Lung Neoplasms; Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Lung Cancer: The Idylla EGFR Mutation Test, performed on the BioCartis Idylla System, is an in vitro diagnostic test for the qualitative detection of exon mutations. One of the biggest challenges in oncology biomarker testing is the ability to obtain samples of sufficient size and quality. This study can help test the BioCartis Idylla System against standard of care (SoC) pathology results from tissue biopsies in the same setting, ultimately being able to diagnose with a fraction of the tissue previously needed.
  Interventions: Diagnostic Test: Idylla EGFR Mutation Test

INTERVENTIONS:
Diagnostic Test: Idylla EGFR Mutation Test — This diagnostic test is performed on the BioCartis Idylla System for qualitative detection of exon mutations.

SUMMARY:
This retrospective, observational study will compare the results of a BioCartis' EGFR mutation test on the Idylla platform with test results from SoC pathology results from tissue biopsies in the same setting. A comparable rapid testing platform for EGFR may serve as a more accessible means to diagnose, and overall, more patients treated successfully with targeted therapies. Up to 150 samples will be tested and compared with existing results.

DETAILED DESCRIPTION:
This study will compare the results of a BioCartis' EGFR mutation test on theIdylla platform with test results from standard of care (SoC) pathology results from tissue biopsies. The Idylla™ EGFR Mutation Test, performed on the BioCartis Idylla™ System, is an in vitro diagnostic test for the qualitative detection of exon 18, exon 20, and exon 21 mutations. Additionally, exon 19 deletions and exon 20 insertions in the EGFR oncogene. A rapid testing platform for EGFR may serve as a more accessible means to diagnose, and overall, more patients treated successfully with targeted therapies.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with primary lung cancer
* Data from primary diagnosis must be included in pathology report or data entry.
* Detailed pathology report included for all samples

Exclusion Criteria:

* Limited or no tissue available
* Only tissue available is from fine needle aspiration
* Tissue blocks older than 5 years old

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Target population is patients diagnosed with primary lung cancer and potentially have known EGFR mutation status.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2021-08 (Estimated); Primary Completion 2022-12 (Estimated); Study Completion 2023-01 (Estimated)

PRIMARY OUTCOMES:
Idylla EGFR Mutation Test | Retrospective tissue samples no longer than 5 years old
  The primary outcome measured is if the Idylla EGFR Mutation Test is a possible alternative to diagnose EGFR mutation status in tissue samples.

CONTACTS AND LOCATIONS:
Overall Officials: Anthony Magliocco, MD, Principal Investigator — CEO and Founder
Locations (1):
- 6555 Sanger Rd, Suite 260, Orlando, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Company Website — https://www.proteanbiodx.com/